CLINICAL TRIAL: NCT05622890
Title: A Single-arm, Phase III Clinical Trial of IMGN853 in Chinese Adult Patients With Platinum-resistant, Advanced High-grade Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer With High Expression of Folate Receptor-α
Brief Title: A Single-arm Clinical Trial of IMGN853 in Chinese Adult Patients With Platinum-resistant, Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-301; CTR20220190 (Registry Identifier: http://www.chinadrugtrials.org.cn/index.html)
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum resistant; Folate-receptor alpha expression; Phase 3; Antibody-drug conjugate; mirvetuximab soravtansine; IMGN853; Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; MIRV; FRα
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): All patients will receive single-agent mirvetuximab soravtansine (MIRV) at 6 mg/kg adjusted ideal body weight (AIBW) administered on Day 1 of every 3-week cycle (Q3W).
  Interventions: Drug: Mirvetuximab Soravtansine

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — Mirvetuximab Soravtansine is an antibody drug conjugate designed to target folate receptor α (FRα). It consists of the humanized anti-FRα mAb M9346A attached via a cleavable disulfide linker to the cytotoxic maytansinoid, DM4.
  Other Names: IMGN853; MIRV

SUMMARY:
This Phase III single-arm study is to evaluate the efficacy and safety of IMGN853 in Chinese adult patients with platinum-resistant high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancers (hereafter referred to as PROC) with high FRα expression.

DETAILED DESCRIPTION:
This is a single-arm, phase III clinical trial of IMGN853 in Chinese adult patients with platinum-resistant, advanced high-grade epithelial ovarian, primary peritoneal or fallopian tube cancer with high expression of folate receptor-α.

The objective of this study is to determine the efficacy of IMGN853 in platinum-resistant ovarian cancer (PROC) patients with high folate receptor alpha (FRα) expression.

A total of 35 patients will be enrolled. All patients must have measurable disease (per Response Evaluation Criteria in Solid Tumors version 1.1, RECIST v1.1) at baseline and be eligible for receiving IMGN853.

All patients will be treated with the IMGN853 monotherapy with a dose at adjusted ideal body weight (AIBW) of 6 mg/kg on Day 1 of every 3-week cycle (Q3W).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥ 18 years of age
2. Patients must have a histopathologically confirmed diagnosis of high-grade serous EOC.
3. Patients must have platinum-resistant disease:

   1. Patients must have had a response (CR or PR) after previous 1 line of platinum-based therapy for at least 4 cycles of treatment, and then progressed between > 3 months and ≤ 6 months after the date for last dose of platinum.
   2. Patients who relapsed after > 6 months since the last platinum-based treatment with at least 4 cycles of one line platinum-based therapy: 1) continued to receive at least 4 cycles of 2 or 3 lines of platinum-based treatment and must have had PD within 6 months from the last dose of platinum; or 2) had PD during treatment with 2 or 3 lines of platinum-containing chemotherapy.

   Note: PD should be calculated from the date of the last dose of platinum-containing therapy to the date of PD indicated by radiographic imaging.

   Note: Patients who are platinum-refractory during 1 line treatment are excluded (see exclusion criterion 3).
4. Patients must have radiological PD on or after the most recent anti-cancer therapy.
5. Patients must be willing to provide the archival tumor tissue slides or undergo low-risk routine medical procedures to collect new biopsy samples for immunohistochemistry (IHC) confirmation of FRα positivity.
6. Per VENTANA FOLR1 (FOLR-2.1) Assay criteria, patient's tumor must be positive for FRα expression by a central laboratory.
7. Patients must have at least one lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically assessed by the investigator).
8. Patients must have received at least 1 but no more than 3 lines of prior systemic anti-cancer therapy, including at least 1 line of therapy containing bevacizumab, and for whom monotherapy is appropriate for the next line of treatment:

   1. Neoadjuvant ± adjuvant is considered as 1 line of therapy;
   2. Maintenance therapy (eg, bevacizumab, PARP inhibitors) will be considered as part of the prior line of therapy (ie, not counted independently);
   3. Therapy changed due to toxicity in the absence of PD will be considered as part of the same line (ie, not counted independently);
   4. Hormonal therapy (except as maintenance therapy) will be considered as a separate line of therapy.
9. Patients must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
10. Patients must have completed prior therapy within the following specified times:

    1. Systemic anti-tumor therapy (the last prior systemic anti-tumor therapy should be at least 5 half-lives or 4 weeks from the initiation of the investigational drug, whichever is shorter);
    2. Focal radiotherapy: previous focal radiotherapy should be at least 2 weeks from the initiation of investigational drug.
11. All toxicities (except alopecia) associated with prior therapy must be stable or resolved (Grade 1 or normal).
12. Any major surgery that a patient has undergone must have been completed at least 4 weeks prior to the first dose of IMGN853 and the postoperative complications of prior surgical treatment have resolved or are stable.
13. Patients must have adequate hematologic, hepatic, and renal functions as defined by the following parameters (without G-CSF [a 20-day drug washout period for long-acting growth factors], human albumin injection and other corrective treatment drugs are not allowed within 14 days before obtaining laboratory test values):

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1,500 μL);
    2. Platelet count ≥ 100 × 10^9/L (100,000/μL) without platelet transfusion in the prior 10 days;
    3. Hemoglobin ≥ 9.0 g/dL without packed red blood cell (PRBC) transfusion in the prior 21 days;
    4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN);
    5. Both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN;
    6. Serum bilirubin ≤ 1.5 × ULN (patients with Gilbert syndrome may be enrolled if total bilirubin is < 3.0 × ULN);
    7. Serum albumin ≥ 2 g/dL.
14. Patients or their legally authorized representatives must be willing and able to sign the ICF and comply with the requirements of the protocol.
15. Women of child bearing potential (WCBP), defined as a sexually mature woman who have not undergone surgical sterilization or who have not been naturally postmenopausal for at least 12 consecutive months (ie, who have had menses any time in the preceding 12 consecutive months) must agree to use effective contraceptive methods; examples included oral, parenteral, or implantable hormonal contraceptive, intrauterine device, barrier contraceptive with spermicide, partner's latex condom or vasectomy) while on study treatment and for at least 12 weeks after the last dose of investigational drug.
16. WCBP must have a negative pregnancy test within 4 days prior to the first dose of IMGN853.
17. The expected survival of the subject is at least 12 weeks as assessed by the investigator.

Exclusion Criteria:

1. Male patients.
2. Patients with endometrioid carcinoma, clear cell carcinoma, mucinous carcinoma, or sarcoma tissue, mixed tumor containing any of the above histologies, or low grade/borderline ovarian tumor.
3. Patients with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first-line platinum-containing chemotherapy.
4. Patients who have received prior wide-field radiotherapy (RT) with at least 20% of the bone marrow affected.
5. Patients with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE).
6. Patients with active or chronic corneal disorders, history of corneal transplant, or active ocular conditions requiring ongoing treatment/monitoring such as uncontrolled glaucoma, wet age-related macular degeneration requiring treatment with intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilloedema, and /or monocular vision.
7. Patients with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Known acute or chronic active hepatitis B (HBsAg positive and HBV DNA viral load ≥ 2500 copies/mL or > 500 IU/mL, if necessary, patients may receive nucleoside prophylactic anti-hepatitis B virus therapy) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive);
   2. Human immunodeficiency virus (HIV) infection;
   3. Active cytomegalovirus infection;
   4. Any other concurrent infectious disease requiring systematic treatment within 2 weeks prior to the first dose of IMGN853.
8. Patients with a history of multiple sclerosis (MS) or other demyelinating diseases and/or Lambert-Eaton syndrome (paraneoplastic syndrome).
9. Patients with clinically significant cardiac disorders, including but not limited to any of the following:

   1. Myocardial infarction ≤ 6 months prior to the first dose;
   2. Unstable angina pectoris;
   3. Uncontrolled congestive cardiac failure (New York Heart Association classification > II);
   4. Uncontrolled ≥ Grade 3 hypertension (per CTCAE criteria);
   5. Uncontrolled cardiac arrhythmias.
10. Patients with a history of hemorrhagic or ischemic stroke within 6 months prior to signing the ICF.
11. Patients with a history of hepatic cirrhosis (Child-Pugh B or C).
12. Patients with a previous clinical diagnosis of or currently ongoing non-infectious interstitial lung disease (ILD), including noninfectious pneumonitis, lung disorders such as pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pulmonitis, severely impaired lung function, etc.
13. Patients requiring folic acid-containing supplements (e.g., folate deficiency).
14. Known hypersensitivity to previous monoclonal antibody therapy or maytansinoids, or to the investigational drug and/or any excipients.
15. Pregnant or lactating women.
16. Patients with prior IMGN853 or other FRα-targeted drug therapies.
17. Known active central nervous system (CNS) and/or leptomeningeal metastases. Patients with untreated but asymptomatic brain metastases, or patients who have radiographically documented progression-free status for at least 4 weeks after treatment and do not require hormonal or antiepileptic therapy for at least 2 weeks may be considered for enrollment.
18. Patients with a history of other malignancies within 3 years prior to enrollment.

    Note: patients with tumors with a negligible risk of metastasis or death (e.g., adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible for inclusion.
19. Patients with pleural effusion, pericardial effusion, or ascites that cannot be controlled by drainage or other means, except the small amount of effusion that without clinical symptoms or do not require clinical intervention.
20. Patients who are detained by a court or administrative decision, receiving psychiatric care against their will, adults who are under the protection of law (under tutorship/curatorship), people who are unable to give their consent, and people who are subject to a legal guardianship.
21. Participated in other clinical studies and received their investigational drugs within 4 weeks prior to the first dose.
22. Subject has other serious systemic diseases or other reasons that are not suitable for participation in this clinical study as evaluated by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the BIRC.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 2 years
  The time interval from initial response (CR or PR) assessed by the investigator and the BIRC to progressive disease (PD) assessed by the BIRC
ORR assessed by the investigator | Up to 2 years
  The best response of CR or PR assessed by the investigator.
DOR assessed by the investigator | Up to 2 years
  The time interval from initial response (CR or PR) assessed by the investigator to PD assessed by the investigator
Treatment-emergent adverse events (TEAEs) and Laboratory results,physical examinations, or vital signs | Up to 2 years
  Adverse Events (AE's) will be evaluated according to the NCI CTCAE v5.0. AE's will be coded using the latest Medical Dictionary for Regulatory Activities (MedDRA) version and summarized per system organ class (SOC) and preferred term (PT).
Determination of CA-125 response with GCIG criteria | Up to 2 years
  GCIG CA-125 response rate will be calculated using the CA-125 Response-Evaluable population and its exact 95% CI will be estimated using the Clopper-Pearson method.
PFS assessed by the BIRC | Up to 2 years
  The time interval from the first dose of IMGN853 to radiographic PD or death assessed by the BIRC, whichever occurs first.
PFS assessed by the investigator | Up to 2 years
  The time interval from the first dose of IMGN853 to radiographic PD or death assessed by the investigator, whichever occurs first.
Overall survival (OS) | Up to 2 years
  The time interval from the first dose of IMGN853 to death
Summary statistics of intact ADC, total Ab (TAb), DM4 and S-methyl DM4 concentration data over time | Up to 2 years
  To assess the PK properties of IMGN853 and its key metabolites
Incidence of seroconversion of ADA caused by IMGN853 and its relationship to safety and efficacy | Up to 2 years
  Subjects will be evaluated for anti-drug antibody (ADA) levels. Confirmatory experiments will be conducted for positive samples. ADA titers and neutralizing antibodies (Nabs) will be further determined as appropriate after the confirmation of positivity.

OTHER OUTCOMES:
Relationship between test results using the companion diagnostic reagent from MEDx Translational Medicine (Suzhou) Co., Ltd. and efficacy of IMGN853 and consistency with VENTANA FOLR1 | Up to 2 years
  Samples will be tested by another CDx at same time to certify the consistency with VENTANA FOLR1

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technolog, Wuhan, Hubei
  - Zhongnan Hospital Affiliated to Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shengyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Tumor Hospital, Shanghai, Shanghai Municipality
  - SIMC, Shanghai, Shanghai Municipality
  - People's Hospital of Shanxi province, Xi’an, Shanxi
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - People's Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Tumor Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Zhengzhou University, Henan, Zhengzhou

IPD SHARING:
Plan to Share IPD: No